CLINICAL TRIAL: NCT05441332
Title: Kinematic and Neuromuscular Deficiencies Phenotypes Associated With Patellofemoral Pain Syndrome : a Cross-sectional Interventional Study
Brief Title: Kinematic and Neuromuscular Deficiencies Phenotypes Associated With Patellofemoral Pain Syndrome
Acronym: PHENOPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP211433; 2021-A01928-33 (Other: France : Ministry of Health)
Record Dates: First submitted 2022-06-14; First posted 2022-07-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral pain syndrome; 3D Kinematics; assessment; clinical phenotypes; dynamic deficiencies
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patellofemoral pain syndrome (Experimental): Kinematic and neuromuscular assessment
  Interventions: Other: EOS Radiation; Behavioral: Semi-structured interview

INTERVENTIONS:
Other: EOS Radiation — One EOS exam of lower extremities
  Other Names: EOS X-ray exams
Behavioral: Semi-structured interview — Semi-structured interview to identify factors influencing patient adherence behavior for a sub-group of 15 patients. By phone, between 1 to 3 months after inclusion.

SUMMARY:
The purpose of this study is to describe and compare the kinematic deficiencies specifically associated with each of the 3 main clinical phenotypes of patellofemoral pain syndrome. The prevalence of patellofemoral pain is high with a high rate of chronicity and recurrence and an overrepresentation of young, athletic and female populations. There are multiple classifications of patellofemoral pain syndrome. A pragmatic classification distinguishes 3 main clinical phenotypes of patellofemoral pain syndrome: with objectively displaceable patella, with extra-patellar alignment problems and without alignment problems.

The pathophysiology of patellofemoral pain syndrome is multifactorial involving static and dynamic dysfunctions of the hip, knee and foot, which remain incompletely elucidated to date. The links between the clinical and biomechanical aspects are still unclear and the kinematic and neuromuscular deficiencies associated with the 3 main clinical phenotypes are poorly understood. A validated non-invasive device allows the 3D evaluation of femorotibial rotations during walking.

DETAILED DESCRIPTION:
The diagnostic process is based on clinical examination. The evolution of measuring tools like radios, RMI and kinematics device allows a more precise diagnostic of patellofemoral Pain syndrome. We still don't know what kind of gait parameters could help to categorize the different phenotypes. With a better understanding of these phenotypes the investigators will be able to propose a better personalized rehabilitation.

Patellofemoral pain syndrome is defined as an anterior knee pain in front of and around the patella. The diagnosis of patellofemoral pain syndrome is based on clinical examination and standard imaging.

The pathophysiology of the patellofemoral pain syndrome is multifactorial involving static and dynamic dysfunctions of the hip, knee and foot, which remain incompletely elucidated to date. The prevalence of patellofemoral pain is high with a high rate of chronicity and recurrence and an overrepresentation of young, athletic and female populations. A pragmatic classification distinguishes 3 main clinical phenotypes of patellofemoral pain syndrome: with objectively displaceable patella, with extra-patellar alignment problems and without alignment problems.

The links between the clinic and biomechanics are still unclear and the kinematics and neuromuscular impairments associated with the 3 main clinical phenotypes are poorly understood.

The KneeKG is an optoelectronic kinematic assessment device using non-invasive sensors and dedicated to real-time measurement of 3D femoro-tibial position and rotations. The kinematic, neuro-muscular, postural and proprioceptive assessments will allow us to better understand the pathophysiology of the patellofemoral pain syndrome, to establish a more accurate diagnosis of the disease, and provide a better understanding of its causes.

Several studies have shown that better adherence to exercise is associated with greater benefit in terms of pain and function in chronic pathologies.

Semi-structured interviews will enable the investigators to assess the impact of information derived from kinematic examination of the knees on adherence to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of SDFP :
* Anterior pain of the knee, mechanical, in front of and around the patella noted at more than 3/10 on a simple numerical scale (ligament or meniscal damage, synovial plicae, tendinopathies, apophysitis, neuromas, and osteoarthritis FT are differential diagnoses),
* Pain during any of the following activities: Going up / down stairs, squats, jumps, jogging, sitting, crouching.
* Duration of knee anterior pain greater than 1 month
* Affiliation to a social insurance
* Signature of the consent to participate

Exclusion Criteria:

* Neurological disorders affecting the lower extremities
* Radiographic FT osteoarthritis
* History of surgery or trauma to the lower limb less than 1 year old
* Intra-articular knee infiltration ≤ 2 months
* Cognitive or behavioral problems making it impossible to assess
* Participates in intervention research or is in the exclusion period following a previous research, if applicable
* Unable to speak, read and write French
* Patients under guardianship or curatorship,
* Patients receiving AME (French State Medical aid)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-12-09 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Amplitude of rotation | Day of inclusion (up to 10 days)
  Amplitude of rotation of the femur with respect to the tibia in the bearing phase in the 3 planes of space

SECONDARY OUTCOMES:
Length measures | Day of inclusion (up to 10 days)
  EOS femoro-tibial alignment
Q angle (in degree) | Day of inclusion (up to 10 days)
  EOS femoro-tibial alignment
Varus valgus(in degree) | Day of inclusion (up to 10 days)
  EOS femoro-tibial alignment
Peak torque (N.m) | Day of inclusion (up to 10 days)
  Quadriceps isokinetic strenght
Total work (N.m) | Day of inclusion (up to 10 days)
  Quadriceps isokinetic strenght
Peak torque (N.m) | Day of inclusion (up to 10 days)
  Hamstrings isokinetic strenght
Total work (N.m) | Day of inclusion (up to 10 days)
  Hamstrings isokinetic strenght
Quadriceps/Hamstring ratio : 2 measure/leg | Day of inclusion (up to 10 days)
Peak torque (N.m) | Day of inclusion (up to 10 days)
  Hip abductors static strenght
Average torque (N.m) | Day of inclusion (up to 10 days)
  Hip abductors static strenght
Time for reaching peak (s) | Day of inclusion (up to 10 days)
  Hip abductors static strenght
Time difference in the onset between the m.vastus lateralis and m.vastus medialis contraction in ms | Day of inclusion (up to 10 days)
  Activity of the quadriceps measured. Electromyogram was used to quantify the electric potential of quadriceps and referred to as 'quadriceps muscle EMG activity' throughout
Y test | Day of inclusion (up to 10 days)
  Static and dynamic unipodal balance
Eccentric step-down test | Day of inclusion (up to 10 days)
  Static and dynamic unipodal balance
Lateral step down test | Day of inclusion (up to 10 days)
  Static and dynamic unipodal balance
Unipodal stabilometric evaluation | Day of inclusion (up to 10 days)
  Static and dynamic unipodal balance
Foot posture index | Day of inclusion (up to 10 days)
  Foot static
Navicular drop test | Day of inclusion (up to 10 days)
  Foot static
Ober's test | Day of inclusion (up to 10 days)
  Muscle hypoextensibility. Quadriceps, harmstrings, calves,
Visual Analog Scale | Day of inclusion (up to 10 days)
  Determine pain / No pain = 0, maximal pain =100
Anterior knee pain scale (AKPS) | Day of inclusion (up to 10 days)
  Questionnaire to determine pain / 13 questions, minimum score = 0 point, maximum score = 100 points
12-Item Short Form Survey (SF-12) | Day of inclusion (up to 10 days)
  Quality of life, to determine pain
Semi-structured interview | From month 1 to month 3
  Semi-structured interview for a sub-group of 15 patients identify factors influencing patient adherence behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Marvin COLEMAN, MSc, PhD student, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis - Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided